CLINICAL TRIAL: NCT01011218
Title: Management of Insomnia in Breast Cancer Patients: A Preliminary Pilot Study
Brief Title: Management of Insomnia in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Oxana Palesh, Assistant Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-17323; K07CA132916-01A1 (NIH); 25740 (Other: University of Rochester - old protocol ID); BRS0008 (Other: OnCore)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Insomnia; Fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BBT-I + Armodafinil (Experimental): Two Brief Behavioral Therapy for Insomnia (BBT-I) sessions in person and additional brief BBT-I sessions over the phone.
  Armodafinil 150 mg/day by mouth.
  Interventions: Behavioral: BBT-I; Drug: Armodafinil
- Behavioral placebo + Armodafinil (Experimental): Control behavioral intervention is a sleep hygiene handout completed by participant.
  Armodafinil 150 mg/day by mouth.
  Interventions: Behavioral: Control; Drug: Armodafinil
- BBT-I without Armodafinil (Sham Comparator): Two Brief Behavioral Therapy for Insomnia (BBT-I) sessions in person and additional brief BBT-I sessions over the phone.
  No pharmaceutical intervention.
  Interventions: Behavioral: BBT-I
- Behavioral placebo without Armodafinil (Placebo Comparator): Control behavioral intervention is a sleep hygiene handout completed by participant.
  No pharmaceutical intervention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: BBT-I — Brief Behavioral Intervention for Insomnia (BBT-I): 2 sessions in person and additional brief sessions over the phone
  Other Names: Brief Behavioral Intervention for Insomnia
  Arms: BBT-I + Armodafinil; BBT-I without Armodafinil
Behavioral: Control — Control behavioral intervention is a sleep hygiene handout completed by participant.
  Other Names: Behavioral placebo
  Arms: Behavioral placebo + Armodafinil; Behavioral placebo without Armodafinil
Drug: Armodafinil — 150 mg by mouth. Armodafinil is the enantiopure compound of the eugeroic modafinil (Provigil), containing only the (R)-(-)-enantiomer of the racemic modafinil.
  Other Names: Nuvigil
  Arms: BBT-I + Armodafinil; Behavioral placebo + Armodafinil

SUMMARY:
To provide preliminary data on the effects of brief behavioral therapy for insomnia (BBT-I) on insomnia in breast cancer patients expecting to receive cancer treatment (unspecified).

Participants will be randomized into 4 groups:

* Arm 1: Brief Behavioral Treatment of Insomnia (BBT-I) + Armodafinil 150 mg/day.
* Arm 2: Behavioral therapy for insomnia (CBT-I) + Armodafinil 150 mg/day.
* Arm 3: Brief Behavioral Treatment of Insomnia (BBT-I) without pharmaceutical intervention.
* Arm 4: Behavioral therapy for insomnia (CBT-I) without pharmaceutical intervention.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of Brief Behavioral Treatment of Insomnia (BBT-I) in the treatment of insomnia in humans.

Insomnia is an extraordinarily common problem for cancer patients that is often associated with diminished social and vocational functioning and QOL. It is also likely that insomnia exacerbates other cancer-related symptoms (eg, fatigue, nausea, depressive mood, pain and/or reduced pain tolerance) and thus gives rise to the possibility of additive or multiplicative interactions. It is possible that untreated insomnia in the context of cancer therapy may lead to chronic forms of insomnia in cancer survivors which, in turn, independently confers risk for increased psychiatric and medical morbidity.

Thus, insomnia, by itself, is a significant problem that requires better understanding in order that its high prevalence can be reduced.

Developing interventions that might prevent onset of insomnia in breast cancer patients is vital.

ELIGIBILITY:
INCLUSION CRITERIA

* Be scheduled for cancer treatment with chemotherapy or biologics (prior chemotherapy and/or diagnosis of metastatic breast are allowed)
* Have at least 6 weeks of treatment remaining
* ≥ 21 years old
* Able to understand written and spoken English
* Able to swallow medication (until amendment omitting armodafinil treatment)
* Score of 3+ on the Sleep Disruption Evaluation form, OR a score of 8+ on Insomnia Severity Index (ISI)

EXCLUSION CRITERIA

* Prior treatment with armodafinil or modafinil (until amendment omitting armodafinil treatment)
* Prior treatment with psycho-stimulant medication within the past 28 days (until amendment omitting armodafinil treatment)
* Prior treatment with antiseizure medications (until amendment omitting armodafinil treatment)
* Has continuously taken sleep medication daily for the last 28 days (until amendment omitting armodafinil treatment)
* History (self-reported) of unstable medical or psychiatric illness (within the last 5 years)
* History of uncontrolled, cardiac disease, hypertension, severe headaches, glaucoma, or seizures (until amendment omitting armodafinil treatment)
* Pregnant or nursing
* History of substance abuse or meet criteria for current alcohol abuse or dependence
* History (self-reported) of chronic, preexisting insomnia, sleep apnea, or restless leg syndrome (RLS)
* Severe hepatic impairment (until amendment omitting armodafinil treatment)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oxana RG Palesh, PhD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811

RESULTS

PARTICIPANT FLOW:
Groups:
- BBT-I + Armodafinil: Two Brief Behavioral Therapy for Insomnia (BBT-I) sessions in person and additional brief BBT-I sessions over the phone.
  Armodafinil 150 mg/day by mouth.
  BBT-I: Brief Behavioral Intervention for Insomnia (BBT-I): 2 sessions in person and additional brief sessions over the phone
  Armodafinil: 150 mg by mouth. Armodafinil is the enantiopure compound of the eugeroic modafinil (Provigil), containing only the (R)-(-)-enantiomer of the racemic modafinil.
- Behavioral Placebo + Armodafinil: Control behavioral intervention is a sleep hygiene handout completed by participant.
  Armodafinil 150 mg/day by mouth.
  Control: Control behavioral intervention is a sleep hygiene handout completed by participant.
  Armodafinil: 150 mg by mouth. Armodafinil is the enantiopure compound of the eugeroic modafinil (Provigil), containing only the (R)-(-)-enantiomer of the racemic modafinil.
- BBT-I Without Armodafinil: Two Brief Behavioral Therapy for Insomnia (BBT-I) sessions in person and additional brief BBT-I sessions over the phone.
  No pharmaceutical intervention.
  BBT-I: Brief Behavioral Intervention for Insomnia (BBT-I): 2 sessions in person and additional brief sessions over the phone
- Behavioral Placebo Without Armodafinil: Control behavioral intervention is a sleep hygiene handout completed by participant.
  No pharmaceutical intervention.
  Control: Control behavioral intervention is a sleep hygiene handout completed by participant.
Period: Overall Study
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
Started | 9 | 9 | 26 | 26
Completed | 9 | 9 | 26 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil | Total
Number analyzed (Participants) | 9 | 9 | 26 | 26 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 23 | 24 | 65
  >=65 years | 0 | 0 | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (10.5) | 46.7 (9.2) | 51.5 (9.0) | 50.3 (8.6) | 50.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 26 | 26 | 70
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4 | 6 | 14
  Not Hispanic or Latino | 1 | 4 | 17 | 11 | 33
  Unknown or Not Reported | 5 | 4 | 5 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 2
  Black or African American | 0 | 0 | 2 | 1 | 3
  White | 8 | 8 | 14 | 16 | 46
  More than one race | 1 | 1 | 3 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 26 | 26 | 70

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: Insomnia Severity Index (ISI) survey questionnaire is a 7-question survey, with each question having 5 possible answers (none, mild, moderate, severe, or very severe), scored as 0, 1, 2, 3, or 4, respectively. The full range of ISI scores is from 0 to 28. Lower scores are considered good, better, or healthy, and increasingly higher scores are considered to indicate greater insomnia. Clinical interpretation is as follows.
  * 0 to 7 No clinically significant insomnia
  * 8 to14 Subthreshold insomnia
  * 15 to 21 Clinical insomnia (moderate severity)
  * 22 to 28 Clinical insomnia (severe)
  ISI survey was conducted at baseline, 3 weeks, 6 weeks, 10 weeks, and 32 weeks. The outcome is reported as the mean ISI score with standard deviation.
Time Frame: up to 32 Weeks
Population: After baseline, it was not uncommon for participants to not contribute data for every time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
Number analyzed (Participants) | 9 | 9 | 26 | 26
units on a scale
  Baseline | 16.3 (7.4) | 14.6 (6.3) | 13.5 (5.2) | 12.1 (5.4)
  3 Weeks: number analyzed (Participants) | 2 | 9 | 23 | 22
  3 Weeks | 13.0 (7.1) | 10.8 (6.5) | 11.4 (7.1) | 12.3 (4.9)
  6 Weeks: number analyzed (Participants) | 6 | 9 | 25 | 24
  6 Weeks | 9 (6.1) | 10 (6.9) | 8.0 (5.7) | 10.5 (6.5)
  10 Weeks: number analyzed (Participants) | 4 | 9 | 24 | 23
  10 Weeks | 6.0 (3.6) | 8.3 (5.6) | 7.8 (4.5) | 10.6 (6.2)
  32 Weeks: number analyzed (Participants) | 1 | 9 | 14 | 16
  32 Weeks | 3.0 (NA) — Cannot generate standard deviation on single value. | 7.6 (4.4) | 7.0 (4.6) | 8.1 (6.3)

2. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) survey questionnaire is a 13-question subset of the 41-question Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire, with each question having 5 possible answers (not at all; a little bit; somewhat; quite a bit; very much), scored as 0, 1, 2, 3, or 4, respectively. The full range of FACIT-Fatigue scores is from 0 to 52. Higher scores are considered good, better, or healthy, and increasingly lower scores are considered to indicate greater fatigue.
  The FACIT-Fatigue survey was conducted at baseline, 3 weeks, 6 weeks, 10 weeks, and 32 weeks. The outcome is reported as the mean with standard deviation.
Time Frame: up to 32 Weeks
Population: After baseline, it was not uncommon for participants to not contribute data for every time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
Number analyzed (Participants) | 9 | 9 | 26 | 26
units on a scale
  Baseline | 27.2 (27.3) | 29.1 (8.2) | 29.1 (12.2) | 30.3 (11.5)
  3 Weeks: number analyzed (Participants) | 6 | 9 | 25 | 25
  3 Weeks | 33.5 (12.5) | 29.6 (10.2) | 29.4 (11.3) | 31.0 (11.5)
  6 Weeks: number analyzed (Participants) | 6 | 9 | 25 | 24
  6 Weeks | 32.5 (10.6) | 33.7 (11.4) | 33.1 (12.4) | 34.2 (11.7)
  10 Weeks: number analyzed (Participants) | 4 | 8 | 24 | 23
  10 Weeks | 41.5 (10.0) | 34.2 (12.7) | 33.2 (11.5) | 34.5 (13.8)
  32 Weeks: number analyzed (Participants) | 1 | 5 | 14 | 16
  32 Weeks | 51 (NA) — Standard deviation cannot be generated from a single value. | 35.8 (4.32) | 37.9 (11.9) | 35.9 (10.8)

3. Other Pre Specified Outcome: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)
Description: The full Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) survey questionnaire is a 41-question survey, with each question having 5 possible answers (not at all; a little bit; somewhat; quite a bit; very much), scored as 0, 1, 2, 3, or 4, respectively. The full range of scores is from 0 to 164. Higher scores are considered good, better, or healthy, and increasingly lower scores are considered to indicate greater fatigue.
  The FACIT-F survey was conducted at baseline, 3 weeks, 6 weeks, 10 weeks, and 32 weeks. The outcome is reported as the mean with standard deviation.
Time Frame: up to 32 Weeks
Population: After baseline, it was not uncommon for participants to not contribute data for every time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
Number analyzed (Participants) | 9 | 9 | 26 | 26
units on a scale
  Baseline | 99.3 (32.0) | 101.2 (21.6) | 100.0 (26.2) | 103.0 (24.4)
  3 Weeks: number analyzed (Participants) | 6 | 9 | 26 | 25
  3 Weeks | 109.8 (25.8) | 99.2 (26.8) | 101.8 (27.3) | 103.3 (29.5)
  6 Weeks: number analyzed (Participants) | 6 | 9 | 26 | 24
  6 Weeks | 110.8 (24.1) | 106.3 (25.8) | 106.4 (31.6) | 108.1 (26.6)
  10 Weeks: number analyzed (Participants) | 4 | 9 | 26 | 23
  10 Weeks | 125.5 (21.6) | 111.2 (29.6) | 107.3 (26.9) | 107.9 (32.0)
  32 Weeks: number analyzed (Participants) | 1 | 9 | 26 | 16
  32 Weeks | 155 (NA) — Standard deviation cannot be generated from a single value. | 118.2 (11.9) | 118.1 (29.2) | 116.4 (23.4)

4. Other Pre Specified Outcome: Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory (BFI) survey questionnaire is a 9-question survey, with each question having 11 possible answers ("No fatigue" to "As bad as you can imagine"), scored from 0 to 10, with each patient's overall BFI score being the mean of the values from each question (overall range 0 to 10). Lower scores are considered good, better, or healthy, and increasingly higher scores are considered to indicate greater fatigue.
  The BFI survey was conducted at baseline, 3 weeks, 6 weeks, 10 weeks, and 32 weeks. The outcome is reported as the mean of the overall BFI scores with standard deviation.
Time Frame: up to 32 Weeks
Population: After baseline, it was not uncommon for participants to not contribute data for every time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
Number analyzed (Participants) | 9 | 9 | 26 | 26
units on a scale
  Baseline | 5.5 (2.6) | 5.2 (2.0) | 4.4 (2.7) | 4.1 (2.4)
  3 Weeks: number analyzed (Participants) | 6 | 9 | 25 | 25
  3 Weeks | 2.8 (1.9) | 4.2 (2.5) | 4.4 (2.8) | 4.0 (2.5)
  6 Weeks: number analyzed (Participants) | 6 | 9 | 25 | 24
  6 Weeks | 4.0 (2.5) | 3.8 (2.5) | 3.0 (2.4) | 3.4 (2.3)
  10 Weeks: number analyzed (Participants) | 4 | 9 | 24 | 23
  10 Weeks | 2.5 (2.2) | 3.1 (2.2) | 3.1 (2.2) | 3.4 (2.6)
  32 Weeks: number analyzed (Participants) | 1 | 9 | 14 | 16
  32 Weeks | 1.0 (NA) — Standard deviation cannot be generated from a single value. | 3.6 (2.0) | 2.7 (2.3) | 3.6 (2.6)

ADVERSE EVENTS:
Arm/Group | BBT-I + Armodafinil | Behavioral Placebo + Armodafinil | BBT-I Without Armodafinil | Behavioral Placebo Without Armodafinil
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/9 | 1/26 | 1/26
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/9 | 1/26 | 1/26
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 5/26 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BBT-I + Armodafinil (N=9) | Behavioral Placebo + Armodafinil (N=9) | BBT-I Without Armodafinil (N=26) | Behavioral Placebo Without Armodafinil (N=26)
Pain, bone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death, not otherwise specified (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BBT-I + Armodafinil (N=9) | Behavioral Placebo + Armodafinil (N=9) | BBT-I Without Armodafinil (N=26) | Behavioral Placebo Without Armodafinil (N=26)
Heart rate increased (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pain, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, breast (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection, bronchial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection, upper respiratory (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain, sinus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No